CLINICAL TRIAL: NCT04473560
Title: Continuous Aspiration Thrombectomy in High and Intermediate-high Risk Pulmonary Embolism Patients
Brief Title: Catheter-directed Thrombectomy in High and Intermediate-high Risk Pulmonary Embolism
Acronym: CATH-PE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aleksander Araszkiewicz, Associate Professor of Medicine, Poznan University of Medical Sciences
Other Study IDs: 879/19
Record Dates: First submitted 2020-07-06; First posted 2020-07-16 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pulmonary Embolism With Acute Cor Pulmonale
Keywords: pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Catheter-directed thrombectomy group: Patients with acute pulmonary embolism treated with catheter-directed thrombectomy along with anticoagulation therapy
  Interventions: Device: Catheter-directed thrombectomy
- No catheter-directed thrombectomy group: Patients with acute pulmonary embolism treated with anticoagulation therapy alone

INTERVENTIONS:
Device: Catheter-directed thrombectomy — Using common femoral venous access the pigtail diagnostic catheter will be placed into the main pulmonary artery and an initial pulmonary angiogram will be performed to demonstrate the location and extent of thrombi in pulmonary arteries. Then pulmonary arterial pressures will be measured. Subsequently an Indigo catheter (Penumbra, Alameda, California) will be placed and a direct-aspiration first-pass technique will be performed purposefully to attach a large thrombus to the catheter tip by suction and then pull it out through the sheath. The decision to terminate the intervention will be at operator's discretion after careful evaluation of hemodynamic parameters (restoration of the systolic blood pressure≥100 mmHg, heart rate <100/min), improvement of arterial blood saturation≥ 92%, practicable clot burden reduction and total amount of aspirated blood (no more than 300 ml).
  Groups: Catheter-directed thrombectomy group

SUMMARY:
Pulmonary embolism is one of the leading causes of cardiovascular death. Pulmonary embolism may be life-threatening condition with an estimated 30-day mortality rate about 10-30%. In high-risk pulmonary embolism, systemic thrombolysis is indicated, whereas recent development of interventional cardiology has made catheter-directed techniques an important alternative to thrombolytic therapy. The controversy concerns also risk stratification and treatment in intermediate-high risk pulmonary embolism patients. A significant percentage of intermediate-high risk patients with pulmonary embolism may experience rapid hemodynamic deterioration and then the prognosis in this group is significantly worse. Catheter-directed techniques are aimed to quickly relive obstruction and restore pulmonary blood flow, thus increasing cardiac output and immediately restoring hemodynamic stability.

The scope of this study is to evaluate the safety and feasibility of catheter-directed approaches in high-risk and intermediate-high risk pulmonary embolism patients.

DETAILED DESCRIPTION:
Pulmonary embolism is one of the leading causes of cardiovascular death. Pulmonary embolism may be life-threatening condition with an estimated 30-day mortality rate about 10-30%. In high-risk pulmonary embolism, systemic thrombolysis is indicated, whereas recent development of interventional cardiology has made catheter-directed techniques an important alternative to thrombolytic therapy. The controversy concerns also risk stratification and treatment in intermediate-high risk pulmonary embolism patients. A significant percentage of intermediate-high risk patients with pulmonary embolism may experience rapid hemodynamic deterioration and then the prognosis in this group is significantly worse. Catheter-directed techniques are aimed to quickly relive obstruction and restore pulmonary blood flow, thus increasing cardiac output and immediately restoring hemodynamic stability.

The scope of this study is to evaluate the safety and feasibility of catheter-directed approaches in high-risk and intermediate-high risk pulmonary embolism patients.

The primary data recorded include details of each patient's clinical status, co-morbidities with the Charlson Comorbidity Index, the implemented catheter-directed therapy, the results of additional studies (lab tests results, electrocardiogram, imaging studies), and the outcome. The study endpoints comprise technical success, clinically relevant procedure-related complications or bleeding events, classified according to the Valve Academic Research Consortium-2 guidelines criteria.

Collecting the fore mentioned data allows for clinicians to better manage the pulmonary embolism patients with increased mortality risk.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms and presentation consistent with pulmonary embolism (PE).
2. PE symptoms duration ≤ 14 days.
3. High risk PE patients with absolute contraindications to systemic thrombolysis or its failure (refractory circulatory collapse) not eligible for surgical embolectomy.
4. Intermediate-high risk PE patients with right ventricle dysfunction confirmed by computed tomography pulmonary angiography or transthoracic echocardiography and elevated troponin level with concomitant at least one of below criterium for minimum 24 hours:

   1. Systolic blood pressure > 90 mmHg and ≤ 100 mmHg
   2. Heart rate ≥ 110/min,
   3. Arterial blood saturation <90% during spontaneous breathing (atm)
5. Intermediate-high risk PE patients with right ventricle dysfunction confirmed by computed tomography pulmonary angiography or transthoracic echocardiography and elevated troponin level with sudden occurrence of one or more of the below listed factors:

   1. Systolic blood pressure > 90 mmHg and ≤ 100 mmHg
   2. Heart rate≥ 110/min,
   3. Arterial blood saturation <90% during spontaneous breathing (atm)

Exclusion Criteria:

1. Pregnancy.
2. Refusal to sign the informed consent form.
3. Presence of intracardiac thrombus.
4. Diagnosed thrombophilia.
5. Severe thrombocytopenia (platelets count below 20 000 µL).
6. History of severe or chronic pulmonary hypertension.
7. Serum creatinine level higher than 1.8 mg/dl.
8. Known serious and uncontrolled sensitivity to radiographic agents.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized due to high risk or intermediate-high risk pulmonary embolism.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of pulmonary arterial pressures | Immediately after catheter-directed thrombectomy procedure
  Incidence of the reduction of systolic and mean pulmonary arterial pressures (mmHg) more than 10% immediately after CDT procedure.
Reduction of vascular obstruction | Immediately after catheter-directed thrombectomy procedure
  Incidence of the at least 50% reduction of vascular obstruction in the angiography assessed with Miller Index score
Clinical improvement during catheter-directed thrombectomy (CDT) procedure | Immediately after catheter-directed thrombectomy procedure
  Incidence of arterial blood saturation increase >92%
Ventricular strain reduction | 24 hours after catheter-directed thrombectomy
  Rate of right ventricular strain reduction (right ventricle/left ventricle ratio assessment) in echocardiography 24 hours after the CDT.
Early mortality rate from pulmonary embolism | 24 hours after catheter-directed thrombectomy
  Number of patients who died from pulmonary embolism (right heart failure) during the first 24 hours after CDT.

SECONDARY OUTCOMES:
Total mortality rate from pulmonary embolism | 3 months after catheter-directed thrombectomy
  1. Number of patients who died from pulmonary embolism (right heart failure)
Bleeding events incidence | 3 months after catheter-directed thrombectomy
  Incidence of major bleedings assessed using The Valve Academic Research Consortium-2 criteria
Adverse events incidence | 3 months after catheter-directed thrombectomy
  Incidence of pulmonary vascular injury assessed on angiography

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Araszkiewicz, Assoc. Prof., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Greaterpoland, Poland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this study, after deidentification (text, figures, tables and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning just after study results publication and ending 24 months following study results publication
Access Criteria: Investigators who provide a methodologically sound proposal. Proposals should be submitted to aaraszkiewicz@ump.edu.pl